CLINICAL TRIAL: NCT02080182
Title: Study of the Effect of Acetylcysteine on Inflammation Biomarkers in Pediatric Acute Pyelonephritis.
Brief Title: Effect of Acetylcysteine in Pediatric Acute Pyelonephritis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jamshid Salamzadeh, PhD, Clinical Pharmacist, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAC1165
Record Dates: First submitted 2014-02-28; First posted 2014-03-06 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Pyelonephritis
Keywords: Acute Pyelonephritis; Acetylcysteine; Pediatric
MeSH Terms: conditions — Pyelonephritis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetylcysteine (Active Comparator): Effervescent tablet of acetylcysteine 600 mg dosing according to weight, until 5 days. Dose for patients more than 30 kg: 1.5 tablet daily 8.5-30 kg: 1 tablet daily less than 8.5 kg: 70 mg/kg
  Interventions: Drug: Acetylcysteine
- Placebo (Placebo Comparator): Placebo effervescent tablet of acetylcysteine 600 mg dosing according to weight, until 5 days. Dose for patients more than 30 kg: 1.5 tablet daily 8.5-30 kg: 1 tablet daily: more than 30 kg: 1.5 tablet daily 8.5-30 kg: 1 tablet daily less than 8.5 kg: 70 mg/kg
  Interventions: Drug: placebo acetylcysteine

INTERVENTIONS:
Drug: Acetylcysteine
  Arms: Acetylcysteine
Drug: placebo acetylcysteine
  Arms: Placebo

SUMMARY:
In different studies, it has been shown that "antioxidant" utilization has favorable therapeutic effects not only on control of acute symptoms but also on prevention of delayed problems from acute and chronic pyelonephritis.

According to the efficacy of acetylcysteine as a potent antioxidant, safety of this drug and side effects of similar or either less than placebo, this study was designed to evaluate the efficacy of this drug on inflammatory biomarkers of pediatric acute pyelonephritis. It is a triple-blind placebo controlled study on a population of 64 patients 1-16 years old that have "definite" or "probable" diagnosis of acute pyelonephritis in "Mofid" hospital.

After randomization, patients will be given acetylcysteine or placebo with dosing according to their weight. Results of treatment are evaluated according to serum procalcitonin, C reactive protein and leukocyte count before drug prescription (baseline) and 5 days after drug prescription. Side effects are also recorded in both groups. Patients will be receiving their routine antimicrobial drugs in addition to acetylcysteine.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 1 and 16
* Having the diagnosis of "definite" or "probable" urinary tract infection according to guidelines of "pediatric infectious disease research center

Exclusion Criteria:

* Patients younger than 1 or older than 16 years old
* Patients without the diagnosis of "definite" or "probable" urinary tract infection according to guidelines of "pediatric infectious disease research center"
* Patients with acute/ chronic infectious or inflammatory diseases other than pyelonephritis.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Serum procalcitonin | Change from baseline serum procalcitonin at 5 days

SECONDARY OUTCOMES:
Serum C Reactive Protein | Change from baseline serum C Reactive Protein at 5 days
Leukocyte count | Change from baseline leukocyte count at 5 days
Probable adverse effects (nausea, vomiting, bad tasting, stomatitis, ...) | Participants will be followed for the duration of hospital stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Infections Research Center, Tehran, Tehran Province, Iran